CLINICAL TRIAL: NCT02936661
Title: Tranexamic Acid for Preventing Postpartum Hemorrhage After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ShanghaiFMIH-TXA1
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Postpartum Hemorrhage， Cesarean Section
Keywords: postpartum hemorrhage， cesarean section， tranexamic acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental): Tranexamic acid 1 g（10ml） IV in 2 minutes after the baby delivered during ceasarean section
  Interventions: Drug: Tranexamic Acid
- placebo (Placebo Comparator): NS 10ml IV in 2 minutes after the baby delivered during ceasarean section
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: Placebo
  Arms: placebo

SUMMARY:
It is a multicenter randomized, double-blind and placebo-controlled trial. Totally 6500 women to delivery by cesarean section will be recruited in this study. In addition to routinely oxytocin, the women in study group will receive TXA 1 g in 2 minutes after they delivered their babies, and those in control group will receive placebo. The incidence of postpartum hemorrhage, the amount of bleeding, as well as the side effects will be observed.

ELIGIBILITY:
Inclusion Criteria:

* gestational week more than 37;
* to delivery by cesarean section;
* informed consent form signed

Exclusion Criteria:

* Any known renal or liver disorders
* History of venous or arterial thrombosis
* Any disease or history tend to increase thrombosis: opertion in 1 month; active smoker.
* Do cesarean section because of active bleeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6700 (Estimated)
Dates: Start 2017-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
postpartum hemorrhage | 24h after the cesarean section

SECONDARY OUTCOMES:
the amount of postpartum bleeding | 24h after the cesarean section

IPD SHARING:
Plan to Share IPD: Undecided